CLINICAL TRIAL: NCT02909127
Title: The Development of the Pediatric Eating Assessment Tool (PEDI-EAT-10)
Brief Title: The Pediatric Eating Assessment Tool
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, PT, PhD, Hacettepe University
Other Study IDs: PEDI-EAT-10
Record Dates: First submitted 2016-08-19; First posted 2016-09-21 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
Keywords: deglutition; deglutition disorders; pediatric dysphagia; swallowing
MeSH Terms: conditions — Cerebral Palsy; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cerebral palsied children: The inclusion criteria are age above 18 months, fed orally, referred due to parent complaints about their child's swallowing function and not admitted a swallowing center before. Swallowing evaluation will be performed. The Functional Independence Measure and PEDI-EAT-10 will be filled.
  Interventions: Other: SWALLOWING EVALUATION; Other: The Functional Independence Measure; Other: The PEDI-EAT-10
- Healthy children: Healthy children above the age of 18 months with no medical history of voice, swallowing, reflux, airway, neurologic, rheumatologic, or neoplastic disorders will be included for normative data generation. The PEDI-EAT-10 will be filled.
  Interventions: Other: The PEDI-EAT-10

INTERVENTIONS:
Other: SWALLOWING EVALUATION — Swallowing function of the CP patients will be imaged and recorded with Videofluoroscopic Swallowing Study (VFSS). The oral cavity, pharynx, larynx and just below the upper esophageal sphincter are visible. 3 trials of 3 ml of liquids will be used and the worst score will be considered for calculation. The Penetration-Aspiration Scale (PAS) will be used to assess dysphagia severity. The PAS is an ordinal scale consisting of eight scores. Scores are determined primarily by the depth to which material passes in the airway and by whether or not material entering the airway is expelled.
  Groups: Cerebral palsied children
Other: The Functional Independence Measure — The Functional Independence Measure for Children (Wee-FIM) will be used to assess the functional independence level of the CP children. The Wee-FIM is developed to emphasize habilitative and developmental aspects of children with special health care needs, genetic disorders, developmental disabilities, and acquired disabilities.
  Groups: Cerebral palsied children
Other: The PEDI-EAT-10 — The PEDI-EAT-10 will also be administered.

SUMMARY:
There is no dysphagia spesific and patient/parent centered outcome instrument in the pediatric population. The purpose of this investigation is to develop the Pediatric version of the Eating Assessment Tool (PEDI-EAT-10) and investigate its validity and reliability.

DETAILED DESCRIPTION:
The evaluation of pediatric swallowing disorders includes clinical and instrumental techniques. The clinical evaluation is important for clinical decision-making and to assess the need for an instrumental evaluation of swallowing. A recent systematic review suggested that the currently available non-instrumental assessments for clinicians to evaluate swallowing and feeding function in the pediatric population have wide variations in design, assessment domains, and target groups. It was concluded that there is a significant need for standardized assessment tools with good psychometric properties in the pediatric population. The existing instruments measure the presence or absence and frequency of challenges related to eating/feeding problems in pediatrics, they do not comprehensively measure oropharyngeal phase swallowing problems or do not reflect the severity of oropharyngeal dysphagia symptoms. The 10-item Eating Assessment Tool (EAT-10), which was designed for adult patients, is a good model for this current research. It has proven highly successful in quantifying initial dysphagia symptom severity and in monitoring treatment efficacy in a vast array of dysphagia etiologies. Although the EAT-10 is a symptom survey, it has been able to predict objective evidence of swallowing dysfunction. There is no dysphagia spesific and patient/parent centered outcome instrument in the pediatric population such as the EAT-10. The purpose of this investigation is to develop the Pediatric version of the Eating Assessment Tool (PEDI-EAT-10) and investigate its validity and reliability.

ELIGIBILITY:
The inclusion criteria are:

* Age above 18 months,
* Fed orally,
* Referred due to parent complaints about their child's swallowing function,
* Not admitted a swallowing center before.

The exclusion criteria are:

* Age below 18 months,
* Fed nonorally,
* No parent complaints about their child's swallowing function,
* Admitted a swallowing center before.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children with spastic cerebral palsy (CP) will be included to test internal consisteny, test-retest reliability and criterion validity.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Development of the scale steps | 10 days
  A comprehensive pediatric dysphagia literature review and the validated items from the other scales will be used to create the items of the PEDI-EAT-10. The PEDI-EAT-10 was designed as a parent-report measure of dysphagia symptom severity. Content validity will also be investigated because it is the first stage of instrument development. An expert panel with Delphi rounds will be convened to determine the initial content validity. The experts will be scored each item of the scale as ''necessary'', ''insufficent'' or ''unnecessary'' and the content validity index (CVI) will be calculated.

SECONDARY OUTCOMES:
Investigation of the psychometric properties of the scale | 6 MONTHS
  The PEDI-EAT-10 will be administered to the primary feeders of the CP children on two separate occasions separated by at least 48 hours to evaluate test-retest reliability. The criterion-related validity of the PEDI-EAT-10 will be assessed by the correlation between the PEDI-EAT-10 and swallowing evaluation results.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lefton-Greif MA. Pediatric dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):837-51, ix. doi: 10.1016/j.pmr.2008.05.007. PMID 18940644
- [Result] Arvedson JC. Assessment of pediatric dysphagia and feeding disorders: clinical and instrumental approaches. Dev Disabil Res Rev. 2008;14(2):118-27. doi: 10.1002/ddrr.17. PMID 18646015
- [Derived] Serel Arslan S, Kilinc HE, Yasaroglu OF, Demir N, Karaduman AA. The pediatric version of the eating assessment tool-10 has discriminant ability to detect aspiration in children with neurological impairments. Neurogastroenterol Motil. 2018 Nov;30(11):e13432. doi: 10.1111/nmo.13432. Epub 2018 Aug 13. PMID 30101572